CLINICAL TRIAL: NCT06222541
Title: Using Online Food Retail "Nudges" to Promote Healthier Beverage Intake Among Low-Income Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-01038
Record Dates: First submitted 2024-01-16; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Nudge" Web-Based Supermarket (Experimental): Participants will be asked to simulate one grocery shopping trip in a web-based supermarket and to select three unique beverages for their household that their child would drink.
  Participants randomized to the "nudge" web-based supermarket will view beverages in descending order of healthfulness (i.e., the healthiest beverages will appear at the top of the screen), view a store landing page promoting the healthiest beverages with a health message, and be offered healthier swaps for sugary drinks at point-of-selection (i.e., immediately after selecting an item to be added to their shopping cart).
  Interventions: Behavioral: "Nudges" in Web-Based Supermarket
- Standard Web-Based Supermarket (No Intervention): Participants will be asked to simulate one grocery shopping trip in a web-based supermarket and to select three unique beverages for their household that their child would drink.
  Participants randomized to the standard web-based supermarket will not receive any nudges related to health.

INTERVENTIONS:
Behavioral: "Nudges" in Web-Based Supermarket — While shopping in the web-based supermarket, participants assigned to the "nudge" arm will see retail nudges to discourage sugary drink purchases and promote healthier substitutes.
  Arms: "Nudge" Web-Based Supermarket

SUMMARY:
The specific aims of this proposal are to 1) develop online food retail nudges to discourage sugary drink purchases and promote healthier substitutes; 2) examine the impact of online store nudges on purchases of sugary drinks in an online randomized controlled experiment with low-income parents, including Supplemental Nutrition Assistance Program (SNAP) and Women, Infants, and Children (WIC)-participating parents, of children age 1-5 years; and 3) disseminate findings to retailers, including those participating in the SNAP Online Purchasing Pilot.

ELIGIBILITY:
Inclusion Criteria:

For Aim 1, the inclusion criteria are as follows:

* parent (or caregiver) of children ages 1-5 years;
* the ability to read and write in English;
* aged 18 years or older;
* household income at or below 185% of the federal poverty level;
* previously purchased fruit drinks for their children;
* have ever shopped for groceries online in the last 12 months,
* live in the US, and
* have access to a personal computer, laptop, or tablet.

The inclusion criteria for Aim 2 are identical to the inclusion criteria for Aim 1, except the researchers will not aim to recruit exclusively parents who have previously purchased sugary drinks for their children or who have ever shopped for groceries online in the last 12 months.

Exclusion Criteria:

The exclusion criteria for Aim 1 include:

* not parent (or caregiver) of children ages 1-5 years;
* aged <18 years or >99 years;
* lack the ability to read and speak English;
* household income above 185% the federal poverty level;
* have never purchased fruit drinks for their children;
* have never shopped for groceries online in the last 12 months;
* do not live in the US, and;
* do not have access to a personal computer, laptop, or tablet. The exclusion criteria for Aim 2 are identical to the exclusion criteria for Aim 1, except participants who have never purchased sugary drinks for their children and have never shopped for groceries online in the last 12 months will not be excluded.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2241 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Total Calories of Sugary Drinks Purchased during Shopping Activity | Day 1 (Approximately 30 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Pasquale Rummo, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: pasquale.rummo@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to pasquale.rummo@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.